CLINICAL TRIAL: NCT04671420
Title: A Phase 3 Multi-Centre, Randomised, Double-Blind, Parallel-Arm Study to Evaluate the Efficacy and Safety of HLX01 Versus Rituximab (Mabthera®) as First Line Treatment in Patients With Low Tumour Burden Follicular Lymphoma.
Brief Title: Evaluate the Efficacy and Safety of HLX01 Versus Mabthera in Patients With Low Tumour Burden Follicular Lymphoma.
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: sponsor strategy decision
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLX01-FL03
Record Dates: First submitted 2020-03-30; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: CD20-positive Follicular Lymphoma, With Low Tumour Burden
MeSH Terms: interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HLX01 (Experimental)
  Interventions: Drug: HLX01
- EU-sourced rituximab (Mabthera®) (Active Comparator)
  Interventions: Drug: Mabthera®

INTERVENTIONS:
Drug: HLX01 — Patients will receive HLX01 intravenous (IV) infusion once a week for 4 weeks induction treatment (on Days 1, 8, 15, and 22), and then continue to receive maintenance treatment at Weeks 12, 20, 28, 36, and 44.
  Arms: HLX01
Drug: Mabthera® — Patients will receive Mabthera® intravenous (IV) infusion once a week for 4 weeks induction treatment (on Days 1, 8, 15, and 22), and then continue to receive maintenance treatment at Weeks 12, 20, 28, 36, and 44.
  Arms: EU-sourced rituximab (Mabthera®)

SUMMARY:
The study is a Phase 3 multi-centre, randomised, double-blind, parallel-arm study to evaluate the efficacy and safety of HLX01 versus European Union (EU)-sourced Mabthera® as first line treatment in patients with low tumour burden FL.

The study will consist of a Screening Period (up to 42 days), Treatment Period (Week 1 to Week 44/Month 11), and End of Study (EOS; Month 12 Visit). Approximately 212 patients (106 in each treatment group) will be enrolled.

Utilising a 1-sided 97.5% CI for the risk difference, a reference proportion of 83.2% for Mabthera®, delta for non-inferiority of -17%, and assuming a true difference of 1%, a sample size of 106 patients per arm (212 total) provides approximately 85% power to show non-inferiority of HLX01 to Mabthera® on a primary endpoint of risk difference in ORR up to Week 28. No dropout is included, as all patients will either have data provided for ORR (based on best response), or will be classed as non-responder.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent before any study-related activities
2. ≥ 18 years of age
3. Histologically-confirmed, stage II to IV NHL (CD20+ FL of grades 1, 2, or 3a) by World Health Organization classification of lymphoid neoplasms (2016 revision) [11]
4. Low tumour burden according to the GELF criteria
5. The Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
6. Availability of tumour sample within 12 months before start of study drug treatment
7. At least 1 bi-dimensionally measurable nodal lesion >1.5 cm or extranodal lesion >1 cm in its longest diameter by CT scan as defined by the Modified Lugano Response Classification 2014
8. Adequate organ function

Exclusion Criteria:

1. Prior treatment for FL. Patients previously treated with radiotherapy for stage I FL may be eligible provided they have a measurable lesion located outside the radiation field
2. Transformation to high-grade lymphoma
3. Patients with advanced disease that are considered for treatment with combined chemo immunotherapy
4. Presence or history of central nervous system (CNS) lymphoma involvement
5. Treatment with an investigational agent within 28 days of the first dose of study drug infusion
6. Prior treatment with a chimeric antibody, including HLX01 and Mabthera®
7. History of another malignancy within 2 years of screening, with the exception of curatively treated non-melanoma skin cancer, carcinoma in situ of the uterine cervix, breast or bladder, localised prostate cancer stage T1c or less - and provided that the patient remains relapse free
8. Major surgery within 28 days of the first dose of study drug infusion (excluding lymph node biopsy)
9. Known human immunodeficiency virus (HIV) infection (Serological test for HIV should be performed at screen unless prohibited by local regulations)
10. Active and/or severe infections, including any ongoing infection requiring IV anti microbial treatment
11. Have a current diagnosis of active tuberculosis
12. Active HBV and a positive serological test for HBV (except seropositive due to HBV vaccination) or hepatitis C virus (HCV)
13. Ongoing immunosuppressant treatment; corticosteroid treatment exceeding 20 mg/day prednisone or equivalent within 7 days of the first dose of study drug infusion
14. Known hypersensitivity or allergy to the active principle and/or formulations' ingredients; history of severe allergy or anaphylaxis to murine or biologic agents
15. Live or live attenuated vaccine within 28 days of the first dose of study drug infusion
16. History of significant cardiac or vascular disease including, but not limited to: history of stroke, unstable angina, myocardial infarction or ventricular arrhythmia requiring medication or mechanical control within 6 months before randomisation; congestive heart failure according to the New York Heart Association (NYHA) Functional Classification class III or IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | rom the first dose of study drug through Week 28
  Overall Response Rate up to Week 28, defined as the proportion of patients achieving either complete response (CR) or PR as best response from the first dose of study drug through Week 28 as assessed by a blinded independent review committee according to the Modified Lugano Response Classification 2014.

SECONDARY OUTCOMES:
AEs | up to 12 months
  adverse events
SAEs | up to 12 months
  serious adverse events
Immunogenicity | up to 12 months
  ADA and neutralising antibody
Time-to-progression of disease (TTPD) | up to 12 months
  Time-to-progression of disease
PFS | up to 12 months
  progression-free survival
Cmax | up to 12 months
  max blood cocentration
Ctrough | up to 12 months
  trough serum concentration after each dose during induction period and selected doses thereafter

IPD SHARING:
Plan to Share IPD: No